CLINICAL TRIAL: NCT03406702
Title: A Phase 2a, Safety, Tolerability, Pharmacokinetics, and Quantitative EEG Study of CX-8998 in Adolescents and Adults With Idiopathic Generalized Epilepsy With Absence Seizures
Brief Title: CX-8998 for Absence Seizures
Acronym: T-WAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CX-8998-CLN2-002
Record Dates: First submitted 2018-01-02; First posted 2018-01-23 (Actual); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Epilepsy
Keywords: Epilepsy, Idiopathic Generalized Epilepsy, Absence Seizures
MeSH Terms: conditions — Epilepsy; Epilepsy, Idiopathic Generalized; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CX-8998 (Experimental): T-type calcium channel blocker
  Interventions: Drug: CX-8998

INTERVENTIONS:
Drug: CX-8998 — T-type calcium channel blocker

SUMMARY:
This is a Phase 2a, open-label study consisting of a screening period of up to 4 weeks and a 4-dose-titration treatment period to a dose of up to 10 mg twice daily (BID) of CX-8998, followed by a 1-week safety follow-up period after the last dose of study medication.

DETAILED DESCRIPTION:
This is a Phase 2a, open-label study consisting of a screening period of up to 4 weeks and a 4-dose-titration treatment period to a dose of up to 10 mg twice daily (BID) of CX-8998, followed by a 1-week safety follow-up period after the last dose of study medication.

Subjects will participate for a total of up to 9 weeks, including screening, the 4-week treatment period and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) indicating that the subject has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
2. Men or non-pregnant, non-breastfeeding women 16 to 55 years-of-age who are able to read and understand written and spoken local language.
3. Clinical diagnosis of IGE (including, but not limited to, CAE, JAE, juvenile myoclonic epilepsy, or Jeavons syndrome) with absence seizures consistent with the International League against Epilepsy Revised Classification of Seizures (2017).
4. Absence seizures persisting despite standard of care (SOC) treatment, defined as treatment with at least 2 AEDs appropriate for the patient's epilepsy syndrome. SOC failure, per investigator discretion, will be defined as insufficient clinical response or intolerable side effects, which precludes use of the appropriate AED.
5. Observation of at least 3 instances of generalized discharges of approximately 2.5 - 4 Hz lasting ≥2 seconds via 24-hour ambulatory EEG (centrally reviewed), with approximately 75% normal background based on age and medication use per the central EEG reader's discretion. Intermittent focal spikes are allowed.
6. On stable doses of one or more antiepileptic medication(s) for at least 30 days. If a subject is not on medication, adequate documentation justifying lack of therapy may be acceptable for the subject after sponsor review. Ketogenic, modified Atkins diet (MAD), or low glycemic diet with stable carbohydrate ratio for at least 30 days before screening is an acceptable antiepileptic therapy. Vagal nerve stimulation at stable settings (for at least 30 days before screening), without use of the magnet, is also acceptable.
7. Body weight ≥ 45 kg at screening.
8. Subjects with reproductive capability including all males and women of child-bearing potential (WOCBP) must agree to practice continuous abstinence or adequate contraception methods (appropriate double barrier method or oral, patch, implant, or injectable contraception) from as soon as feasible during screening period until at least 30 days after the last dose (i.e., intermittent abstinence based on "rhythm", temperature monitoring, or other means of timing is not acceptable). WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy) or is not post-menopausal. Post-menopausal is defined as amenorrhea ≥ 12 consecutive months without another cause, and a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.
9. Male subjects with a partner of child-bearing potential must be surgically sterilized or be willing to use condoms with spermicide from as soon as feasible during screening period until at least 30 days after the last dose.
10. Able and willing to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
11. Approval by the sponsor medical personnel or delegate as to final eligibility for the study.

Exclusion Criteria:

1. History of surgical intervention for treatment of epilepsy.
2. Additional seizure (clinical and electrographic) types, including, but not limited to, epileptic spasms, generalized tonic seizures, atonic seizures, or focal seizures. Subjects with GTCS or myoclonic seizures are eligible for the study.
3. Inadequately treated psychotic or mood disorder (e.g., schizophrenia, major depression, bipolar disorder).
4. Presence of severe intellectual disability, severe autism spectrum disorder, or severe developmental disorder such that the subject cannot sign the ICF or cannot cooperate with the study procedures.
5. Presence of positive urine drug screen for drugs of abuse, except if this is explained by use of an allowed prescription medicine.
6. Regular use of more than 2 standard drinks of alcohol per day (28 grams of pure alcohol).
7. Hypersensitivity/allergic reaction to other T-type calcium agents, such as (but not limited to) ethosuximide and zonisamide.
8. Use of strong CYP3A4 inhibitors, including prescription or non-prescription drugs or other products (i.e. grapefruit juice), which cannot be discontinued at least 2 weeks prior to Day 1 of dosing and throughout the study (Appendix C).
9. Concurrent illnesses that would be a contraindication to trial participation, including, but not limited to:

   1. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before screening
   2. NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled hypertension
   3. Clinically significant ECG abnormality per the Investigator assessment or any of the following: i) QTcF ≥450 msec (males) or ≥470 msec (females) ii) PR interval ≥250 msec iii) Atrioventricular block of second degree or higher, including Mobitz I iv) Persistent sinus bradycardia ≤ 50 beats per minute; persistent means the bradycardia is present on the first ECG and on one repeat ECG performed on another day v) For other ECG findings (e.g., including, but not necessarily limited to, tachycardia, bundle branch block, frequent ectopic beats, etc.) the Investigator should send a scanned, identity-blinded copy of the ECG tracing to the Study Safety Representative for review.
10. Positive result for HIV, Hepatitis B [indicating ongoing infection], or Hepatitis C at screening or otherwise known ongoing infection with HIV, hepatitis B, or hepatitis C, unless curative therapy completed; for hepatitis C curative therapy is defined as negative PCR for HCV RNA.
11. Significant hepatic (AST/ALT or bilirubin ≥ 2X upper limit of normal) or renal disease (creatinine clearance ≤39 mL/min) at screening.
12. History of alcohol or substance abuse within the last year.
13. A current C-SSRS score of 4 or 5 at screening or history of suicide attempt.
14. Psychological, social, familial, or geographical reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.
15. Any other condition and/or situation that causes the Investigator or Study Safety Representative to deem a subject unsuitable for the study (including, but not limited to, expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures).
16. Treatment with an investigational agent within 30 days prior to the first dose of CX-8998 or planning to receive an investigational agent during the study.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arkansas Epilepsy Program, Little Rock, Arkansas
  - University of Florida, Tampa, Florida
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - NYU Comprehensive Epilepsy Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent a screening period of up to 4 weeks.
Groups:
- CX-8998: Participants underwent a 4-week dose-titration treatment period up to a dose of 10 mg twice daily (BID) of suvecaltamide in the following schedule: Days 1 to 2: 2 mg BID (4 mg/d); Days 3 to 8: 4 mg BID (8 mg/d); Days 9 to 14: 6 mg BID (12 mg/d); Days 15 to 20: 8 mg BID (16 mg/d); Days 21 to 26: 10 mg BID (20 mg/d).
Period: Overall Study
Arm/Group | CX-8998
Started | 7
Completed | 6
Not Completed | 1
Not completed — Missed Day 27 Dosing | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Intent-to-Treat Population.
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF)
Description: Fridericia's Correction Formula (QTCF) is a formula which takes into account the physiologic shortening of the QT interval which occurs as the heart rate increases, permitting comparison of the QT interval across a range of rates.
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: QTcF was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CX-8998
Number analyzed (Participants) | 6
msec | 3.50 (10.213)

2. Primary Outcome: Change From Baseline to End of Treatment in Clinical Alanine Aminotransferase Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in alanine aminotransferase serum chemistry concentration.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical alanine aminotransferase serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
U/L | 17.29 (33.604)

3. Primary Outcome: Change From Baseline to End of Treatment in Clinical Albumin Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in albumin serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical albumin serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
g/L | -0.29 (4.152)

4. Primary Outcome: Change From Baseline to End of Treatment in Clinical Albumin/Globulin Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in albumin/globulin serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical albumin/globulin serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 7
ratio | -0.15 (0.212)

5. Primary Outcome: Change From Baseline to End of Treatment in Clinical Alkaline Phosphatase Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in alkaline phosphatase serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical alkaline phosphatase serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
U/L | 3.14 (10.399)

6. Primary Outcome: Change From Baseline to End of Treatment in Clinical Aspartate Aminotransferase Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in aspartate aminotransferase serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical aspartate aminotransferase serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
U/L | 27.71 (60.810)

7. Primary Outcome: Baseline Clinical Blood Urea Nitrogen/Creatinine Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in BUN/Creatinine serum chemistry.
Time Frame: Baseline (Day 1)
Population: Clinical BUN/Creatinine serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 1
ratio | 12.70 (NA) — Only 1 participant was analyzed so standard deviation could not be calculated for this assessment.

8. Primary Outcome: Change From Baseline to End of Treatment in Clinical Bilirubin Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in bilirubin serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical bilirubin serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
umol/L | -0.55 (2.577)

9. Primary Outcome: Change From Baseline to End of Treatment in Clinical Blood Urea Nitrogen Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in blood urea nitrogen serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical blood urea nitrogen serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
umol/L | 0.23 (1.254)

10. Primary Outcome: Change From Baseline to End of Treatment in Clinical Carbon Dioxide Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in carbon dioxide serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical carbon dioxide serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | 0.43 (2.936)

11. Primary Outcome: Change From Baseline to End of Treatment in Clinical Chloride Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in chloride serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical chloride serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | -0.86 (3.716)

12. Primary Outcome: Change From Baseline to End of Treatment in Clinical Calcium Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in calcium serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical calcium serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | -0.01 (0.109)

13. Primary Outcome: Change From Baseline to End of Treatment in Clinical Cholesterol Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in cholesterol serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical cholesterol serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | 0.60 (0.895)

14. Primary Outcome: Baseline Clinical Cholesterol/HDL-Cholesterol Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in cholesterol/HDL-cholesterol serum chemistry.
Time Frame: Baseline (Day 1)
Population: Clinical cholesterol/HDL-cholesterol serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 1
ratio | 2.40 (NA) — Only 1 participant was analyzed so standard deviation could not be calculated for this assessment.

15. Primary Outcome: Change From Baseline to End of Treatment in Clinical Creatine Kinase Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in creatine kinase serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical creatine kinase serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
U/L | 1174.86 (3110.151)

16. Primary Outcome: Change From Baseline to End of Treatment in Clinical Creatinine Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in creatinine serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical creatinine serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
umol/L | -4.14 (9.737)

17. Primary Outcome: Change From Baseline to End of Treatment in Clinical Globulin Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in globulin serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical globulin serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | CX-8998
Number analyzed (Participants) | 2
g/dL | 0.15 (0.071)

18. Primary Outcome: Baseline Clinical Glomerular Filtration Rate (GFR) Adjusted for Body Surface Area (BSA) Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in glomerular filtration rate adjusted for BSA chemistry.
Time Frame: Baseline (Day 1)
Population: The clinical glomerular filtration rate adjusted for BSA serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: mL/sec/1.73m^2
Arm/Group | CX-8998
Number analyzed (Participants) | 1
mL/sec/1.73m^2 | 1.80 (NA) — Only 1 participant was analyzed so standard deviation could not be calculated for this assessment.

19. Primary Outcome: Change From Baseline to End of Treatment in Clinical Estimated Glomerular Filtration Rate (GFR) Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in GFR serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical GFR serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: mL/sec/1.73m^2
Arm/Group | CX-8998
Number analyzed (Participants) | 7
mL/sec/1.73m^2 | -5.82 (9.691)

20. Primary Outcome: Change From Baseline to End of Treatment in Clinical Glucose Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in glucose serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical glucose serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | -0.14 (0.526)

21. Primary Outcome: Baseline Clinical HDL Cholesterol Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in HDL cholesterol serum chemistry.
Time Frame: Baseline (Day 1)
Population: Clinical HDL-cholesterol serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 1
nmol/L | 1.35 (NA) — Only 1 participant was analyzed so standard deviation could not be calculated for this assessment.

22. Primary Outcome: Baseline Clinical LDL Cholesterol Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in LDL cholesterol serum chemistry.
Time Frame: Baseline (Day 1)
Population: Clinical LDL-cholesterol serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 1
nmol/L | 1.50 (NA) — Only 1 participant was analyzed so standard deviation could not be calculated for this assessment.

23. Primary Outcome: Change From Baseline to End of Treatment in Clinical Lactate Dehydrogenase Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in lactate dehydrogenase serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical lactate dehydrogenase serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
U/L | 53.86 (98.104)

24. Primary Outcome: Change From Baseline to End of Treatment in Clinical Magnesium Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in magnesium serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical magnesium serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | -0.02 (0.077)

25. Primary Outcome: Baseline Clinical Non-HDL Cholesterol Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in non-HDL cholesterol serum chemistry.
Time Frame: Baseline (Day 1)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 1
nmol/L | 1.84 (NA) — Only 1 participant was analyzed so standard deviation could not be calculated for this assessment.

26. Primary Outcome: Change From Baseline to End of Treatment in Clinical Phosphate Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in phosphate serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical phosphate serum chemistry was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
nmol/L | 0.09 (0.163)

27. Primary Outcome: Change From Baseline to End of Treatment in Clinical Potassium Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in potassium serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical potassium serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | 0.34 (0.532)

28. Primary Outcome: Change From Baseline to End of Treatment in Clinical Protein Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in protein serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical protein serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
g/L | 0.29 (3.352)

29. Primary Outcome: Change From Baseline to End of Treatment in Clinical Sodium Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in sodium serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical sodium serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | -0.57 (1.902)

30. Primary Outcome: Change From Baseline to End of Treatment in Clinical Triglycerides Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in triglycerides serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical triglycerides serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | 0.17 (0.659)

31. Primary Outcome: Change From Baseline to End of Treatment in Clinical Urate Serum Chemistry Concentration
Description: Clinical safety laboratory assessment in urate serum chemistry.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical urate serum chemistry was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
umol/L | 8.71 (48.555)

32. Primary Outcome: Change From Baseline to End of Treatment in Basophils Hematology Assessment
Description: Clinical safety laboratory basophils hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical basophils were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | 0.02 (0.029)

33. Primary Outcome: Change From Baseline to End of Treatment in Basophils/Leukocytes Hematology Assessment
Description: Clinical safety laboratory basophils/leukocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical basophils/leukocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 6
ratio | 0.00 (0.004)

34. Primary Outcome: Change From Baseline to End of Treatment in Eosinophils Hematology Assessment
Description: Clinical safety laboratory eosinophils hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical eosinophils were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | 0.02 (0.042)

35. Primary Outcome: Change From Baseline to End of Treatment in Eosinophils/Leukocytes Hematology Assessment
Description: Clinical safety laboratory eosinophils/leukocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical eosinophils/leukocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 6
ratio | 0.00 (0.007)

36. Primary Outcome: Change From Baseline to End of Treatment in Mean Corpuscular Hemoglobin (HGB) Concentration Hematology Assessment
Description: Clinical safety laboratory mean corpuscular HGB concentration hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical mean corpuscular HGB concentration was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 2
nmol/L | 0.00 (1.230)

37. Primary Outcome: Change From Baseline to End of Treatment in Mean Corpuscular Hemoglobin (HGB) Hematology Assessment
Description: Clinical safety laboratory mean corpuscular HGB hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical mean corpuscular HGB was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: fmol
Arm/Group | CX-8998
Number analyzed (Participants) | 2
fmol | -0.04 (0.049)

38. Primary Outcome: Change From Baseline to End of Treatment in Mean Corpuscular Volume Hematology Assessment
Description: Clinical safety laboratory mean corpuscular volume hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical mean corpuscular volume was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | CX-8998
Number analyzed (Participants) | 2
fL | -1.00 (2.828)

39. Primary Outcome: Change From Baseline to End of Treatment in Erythrocytes Hematology Assessment
Description: Clinical safety laboratory erythrocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical erythrocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E12/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E12/L | -0.02 (0.194)

40. Primary Outcome: Change From Baseline to End of Treatment in Erythrocytes Distribution Width Hematology Assessment
Description: Clinical safety laboratory erythrocytes distribution width hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical erythrocytes distribution width was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 2
ratio | 0.00 (0.000)

41. Primary Outcome: Change From Baseline to End of Treatment in Hematocrit Hematology Assessment
Description: Clinical safety laboratory hematocrit hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical hematocrit was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 6
ratio | 0.00 (0.015)

42. Primary Outcome: Change From Baseline to End of Treatment in Hemaglobin Hematology Assessment
Description: Clinical safety laboratory hemaglobin hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Clinical hemoglobin was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
g/L | 1.17 (6.555)

43. Primary Outcome: Change From Baseline to End of Treatment in Leukocytes Hematology Assessment
Description: Clinical safety laboratory leukocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Leukocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | 0.25 (2.228)

44. Primary Outcome: Change From Baseline to End of Treatment in Lymphocytes Hematology Assessment
Description: Clinical safety laboratory lymphocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Lymphocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | -0.17 (0.452)

45. Primary Outcome: Change From Baseline to End of Treatment in Lymphocytes/Leukocytes Hematology Assessment
Description: Clinical safety laboratory lymphocytes/leukocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Lymphocytes/leukocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 6
ratio | -0.02 (0.045)

46. Primary Outcome: Change From Baseline to End of Treatment in Mean Platelet Volume Hematology Assessment
Description: Clinical safety laboratory mean platelet volume hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Mean platelet volume was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | CX-8998
Number analyzed (Participants) | 2
fL | 0.65 (1.202)

47. Primary Outcome: Change From Baseline to End of Treatment in Monocytes Hematology Assessment
Description: Clinical safety laboratory monocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Monocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | 0.01 (0.067)

48. Primary Outcome: Change From Baseline to End of Treatment in Monocytes/Leukocytes Hematology Assessment
Description: Clinical safety laboratory monocytes/leukocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Monocytes/leukocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 6
ratio | 0.00 (0.021)

49. Primary Outcome: Change From Baseline to End of Treatment in Neutrophils Hematology Assessment
Description: Clinical safety laboratory neutrophils hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Neutrophils were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | 0.41 (1.911)

50. Primary Outcome: Change From Baseline to End of Treatment in Neutrophils/Leukocytes Hematology Assessment
Description: Clinical safety laboratory neutrophils/leukocytes hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Neutrophils/leukocytes were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CX-8998
Number analyzed (Participants) | 6
ratio | 0.02 (0.063)

51. Primary Outcome: Change From Baseline to End of Treatment in Platelets Hematology Assessment
Description: Clinical safety laboratory platelets hematology assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Platelets were assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: cellsx10E9/L
Arm/Group | CX-8998
Number analyzed (Participants) | 6
cellsx10E9/L | 10.67 (38.645)

52. Primary Outcome: Baseline to End of Treatment in Bacteria Urinalysis Assessment
Description: Clinical safety laboratory bacteria urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Bacteria urinalysis was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Not seen) | 1
  End of Treatment (Few) | 1

53. Primary Outcome: Baseline to End of Treatment in Urine Bilirubin Urinalysis Assessment
Description: Clinical safety laboratory urine bilirubin urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Urine bilirubin was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Negative) | 4
  End of Treatment (Negative) | 2

54. Primary Outcome: Baseline to End of Treatment in Epithelial Cells Urinalysis Assessment
Description: Clinical safety laboratory epithelial cells urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed. A normal range is 0-10 epithelial cells/high power field (hpf). A worse outcome is >10 epithelial cells.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Epithelial cells were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (0-10) | 1
  End of Treatment (>10) | 1

55. Primary Outcome: Baseline to End of Treatment in Urine Erythrocytes Urinalysis Assessment
Description: Clinical safety laboratory urine erythrocytes urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed. A normal range is 0-2 erythrocytes/high power field (hpf). A better outcome is 0 or "none seen."
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Urine erythrocytes were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (0-2) | 1
  End of Treatment (None seen) | 1

56. Primary Outcome: Baseline to End of Treatment in Urine Glucose Urinalysis Assessment
Description: Clinical safety laboratory urine glucose urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Urine glucose were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Negative) | 4
  End of Treatment (Negative) | 2

57. Primary Outcome: Baseline to End of Treatment in Ketones Urinalysis Assessment
Description: Clinical safety laboratory ketones urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Ketones were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Negative) | 3
  Baseline (Trace) | 1
  End of Treatment (Negative) | 2

58. Primary Outcome: Baseline to End of Treatment in Leukocyte Esterase Urinalysis Assessment
Description: Clinical safety laboratory leukocyte esterase urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed. A normal assessment or better outcome is "negative." An abnormal assessment or worse outcome is a positive assessment (i.e., 2+).
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Leukocyte esterase was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Negative) | 4
  End of Treatment (2+) | 1
  End of Treatment (Negative) | 1

59. Primary Outcome: Baseline to End of Treatment in Urine Leukocytes Urinalysis Assessment
Description: Clinical safety laboratory urine leukocytes urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed. A normal range is 0-5 leukocytes/high power field (hpf). An abnormal assessment or worse outcome is >5 leukocytes/hpf (i.e., 11-30).
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Urine leukocytes were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (0-5) | 1
  End of Treatment (11-30) | 1

60. Primary Outcome: Baseline to End of Treatment in Mucous Threads Urinalysis Assessment
Description: Clinical safety laboratory mucous threads urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Mucous threads were assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Present) | 1
  End of Treatment (Present) | 1

61. Primary Outcome: Baseline to End of Treatment in Nitrite Urinalysis Assessment
Description: Clinical safety laboratory nitrite urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Nitrite was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Negative) | 4
  End of Treatment (Negative) | 2

62. Primary Outcome: Baseline to End of Treatment in Occult Blood Urinalysis Assessment
Description: Clinical safety laboratory occult blood urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed. A normal assessment or better outcome is "negative." An abnormal assessment or worse outcome is a positive assessment (i.e., 2+).
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Occult blood was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (2+) | 1
  Baseline (Negative) | 3
  End of Treatment (Negative) | 2

63. Primary Outcome: Baseline to End of Treatment in Protein Urinalysis Assessment
Description: Clinical safety laboratory protein urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Protein was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Negative) | 4
  End of Treatment (Negative) | 2

64. Primary Outcome: Baseline to End of Treatment in Specific Gravity Urinalysis Assessment
Description: Clinical safety laboratory specific gravity urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed. A normal assessment or better outcome is 1.005-1.030. An abnormal assessment or worse outcome is a value outside of this range.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Specific gravity was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (1.015) | 1
  Baseline (1.019) | 1
  Baseline (1.025) | 1
  Baseline (1.029) | 1
  End of Treatment (1.023) | 1
  End of Treatment (1.024) | 1
  End of Treatment (1.026) | 1

65. Primary Outcome: Baseline to End of Treatment in Specimen Appearance Urinalysis Assessment
Description: Clinical safety laboratory specimen appearance urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Specimen appearance was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Clear) | 4
  End of Treatment (Clear) | 1
  End of Treatment (Cloudy) | 1
  End of Treatment (Turbid) | 1

66. Primary Outcome: Change From Baseline to End of Treatment in Urobilinogen Urinalysis Assessment
Description: Clinical safety laboratory urobilinogen urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Urobilinogen was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | CX-8998
Number analyzed (Participants) | 7
nmol/L | 0.00 (0.000)

67. Primary Outcome: Baseline to End of Treatment in pH Urinalysis Assessment
Description: Clinical safety laboratory pH urinalysis assessment. Shifts from baseline to normal/abnormal status were assessed.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: pH was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (5) | 1
  Baseline (6) | 1
  Baseline (6.6) | 1
  Baseline (7) | 1
  End of Treatment (5) | 1
  End of Treatment (5.5) | 2

68. Primary Outcome: Baseline to End of Treatment in Urine Color Urinalysis Assessment
Description: Clinical safety laboratory urine color urinalysis assessment.
Time Frame: Baseline (Day 1) to end of treatment, or up to 4 weeks post-dose.
Population: Urine color was assessed using the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | CX-8998
Number analyzed (Participants) | 7
Participants
  Baseline (Yellow) | 4
  End of Treatment (Yellow) | 2

69. Primary Outcome: Number (%) of Participants Who Did Not Complete The Study Due to Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events are all adverse events occurring during the treatment period or a pretreatment event that worsens in intensity during the treatment period as assessed by CTCAE v4.0.
Time Frame: Baseline (Day 1) up to Day 26 post-dose, or up to 1 year 3 weeks.
Population: Participants who did not complete the study was assessed using the safety population. The number of participants analyzed varied as participation declined over time.
Measure: Count of Participants; unit: Participants
Groups:
- CX-8998 Days 1 - 2 (4 mg/d): Participants were administered suvecaltamide orally 2mg capsules twice daily (4 mg/d) on Days 1 to 2.
- CX-8998 Days 3 - 8 (8 mg/d): Participants were administered suvecaltamide orally 2- 2mg capsules twice daily (8 mg/d) on Days 3 to 8.
- CX-8998 Days 9 - 14 (12 mg/d): Participants were administered suvecaltamide orally 3- 2mg capsules twice daily (12 mg/d) on Days 9 to 14.
- CX-8998 Days 15 - 20 (16 mg/d): Participants were administered suvecaltamide orally 4-2mg capsules twice daily (16 mg/d) on Days 15 to 20.
- CX-8998 Days 21 - 27 (20 mg/d): Participants were administered suvecaltamide orally 5-2mg capsules twice daily (20 mg/d) on Days 21 to 27.
Arm/Group | CX-8998 Days 1 - 2 (4 mg/d) | CX-8998 Days 3 - 8 (8 mg/d) | CX-8998 Days 9 - 14 (12 mg/d) | CX-8998 Days 15 - 20 (16 mg/d) | CX-8998 Days 21 - 27 (20 mg/d)
Number analyzed (Participants) | 7 | 5 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

70. Primary Outcome: Number (%) of Participants With Adverse Events of Special Interest
Description: An adverse event of special interest is a serious adverse event as defined in Outcome 6. This includes, however is not limited to, increased seizure frequency, new seizure types, worsening of EEG parameters, systemic adverse events based on safety profile as assessed by CTCAE v4.0.
Time Frame: Baseline (Day 1) up to Day 26 post-dose, or up to 1 year 3 weeks.
Population: Participants with adverse events of special interest were assessed using the safety population. The number of participants analyzed varied as participation declined over time.
Measure: Count of Participants; unit: Participants
Groups:
- CX-8998 Days 1 - 2 (4 mg/d): Participants were administered suvecaltamide orally in 2mg capsules twice daily (4 mg/d) on Days 1 to 2.
- CX-8998 Days 3 - 8 (8 mg/d): Participants were administered suvecaltamide orally 2-2mg capsules twice daily (8 mg/d) on Days 3 to 8.
- CX-8998 Days 9 - 14 (12 mg/d): Participants were administered suvecaltamide orally 3-2mg capsules twice daily (12 mg/d) on Days 9 to 14.
Arm/Group | CX-8998 Days 1 - 2 (4 mg/d) | CX-8998 Days 3 - 8 (8 mg/d) | CX-8998 Days 9 - 14 (12 mg/d) | CX-8998 Days 15 - 20 (16 mg/d) | CX-8998 Days 21 - 27 (20 mg/d)
Number analyzed (Participants) | 7 | 5 | 6 | 6 | 6
Participants
  Any Event | 1 | 0 | 0 | 0 | 1
  Seizure | 1 | 0 | 0 | 0 | 1

71. Primary Outcome: Change From Baseline to End of Treatment in Respiration Rate
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: Respiration rate was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | CX-8998
Number analyzed (Participants) | 7
breaths/min | 0.29 (1.380)

72. Primary Outcome: Change From Baseline to End of Treatment in Temperature
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: Temperature was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | CX-8998
Number analyzed (Participants) | 7
celsius | -0.01 (0.430)

73. Primary Outcome: Baseline Weight
Time Frame: Baseline (Day 1)
Population: Weight was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | CX-8998
Number analyzed (Participants) | 7
kg | 82.19 (15.963)

74. Primary Outcome: Change From Baseline to End of Treatment in Pulse
Description: The change from baseline to end of treatment in participants' pulses was assessed. The changes in recumbent pulse, standing pulse, and the change from recumbent to standing pulse are reported. Change from recumbent to standing pulse was measured by the difference in recumbent pulse change and standing pulse change.
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: Pulse was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | CX-8998
Number analyzed (Participants) | 7
bpm
  Recumbent | -9.71 (8.036)
  Standing | -5.57 (6.973)
  Change from Recumbent to Standing | 4.14 (5.956)

75. Primary Outcome: Change From Baseline to End of Treatment in Systolic Blood Pressure
Description: The change from baseline to end of treatment in participants' systolic blood pressure (sbp) was assessed. The changes in recumbent sbp, standing sbp, and the change from recumbent to standing sbp are reported. Change from recumbent to standing sbp was measured by the difference in recumbent sbp change and standing sbp change.
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: Systolic blood pressure was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CX-8998
Number analyzed (Participants) | 7
mmHg
  Recumbent | -3.29 (14.338)
  Standing | -2.86 (12.103)
  Change from Recumbent to Standing | 0.43 (4.962)

76. Primary Outcome: Change From Baseline to End of Treatment in Diastolic Blood Pressure
Description: The change from baseline to end of treatment in participants' diastolic blood pressure (dbp) was assessed. The changes in recumbent dbp, standing dbp, and the change from recumbent to standing dbp are reported. Change from recumbent to standing dbp was measured by the difference in recumbent dbp change and standing dbp change.
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: Diastolic blood pressure was assessed using the safety population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CX-8998
Number analyzed (Participants) | 7
mmHg
  Recumbent | -8.14 (14.916)
  Standing | 1.86 (7.267)
  Change from Recumbent to Standing | 10.00 (8.737)

77. Primary Outcome: Change From Baseline to End of Treatment in QT Interval
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: QT was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CX-8998
Number analyzed (Participants) | 6
msec | -2.67 (12.801)

78. Primary Outcome: Change From Baseline to End of Treatment in QRS Interval
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: QRS interval was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CX-8998
Number analyzed (Participants) | 6
msec | -1.50 (2.811)

79. Primary Outcome: Change From Baseline to End of Treatment in PR Interval
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: PR interval was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CX-8998
Number analyzed (Participants) | 6
msec | -0.17 (7.026)

80. Primary Outcome: Change From Baseline to End of Treatment in Heart Rate
Time Frame: Baseline (Day 1) to end of treatment 1-2 hours post-dose, up to 4 weeks post-dose.
Population: Heart rate was assessed using the safety population. The number of participants varied due to the lack of completion of assessments.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | CX-8998
Number analyzed (Participants) | 6
beats/min | 3.67 (13.866)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day 1 up to Day 26 post-dose, or up to 1 year 3 weeks.
Description: Treatment-emergent adverse events (TEAEs) are all adverse events (AEs) occurring during the treatment period or a pretreatment event that worsens in intensity during the treatment period. The number of participants varied during Days 3-8 due to the lack of completion of assessments.
Arm/Group | CX-8998 Days 1 - 2 (4 mg/d) | CX-8998 Days 3 - 8 (8 mg/d) | CX-8998 Days 9 - 14 (12 mg/d) | CX-8998 Days 15 - 20 (16 mg/d) | CX-8998 Days 21 - 27 (20 mg/d)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/7 | 2/5 | 0/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CX-8998 Days 1 - 2 (4 mg/d) (N=7) | CX-8998 Days 3 - 8 (8 mg/d) (N=5) | CX-8998 Days 9 - 14 (12 mg/d) (N=6) | CX-8998 Days 15 - 20 (16 mg/d) (N=6) | CX-8998 Days 21 - 27 (20 mg/d) (N=6)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Sluggishness (General disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT03406702/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT03406702/SAP_001.pdf